CLINICAL TRIAL: NCT02766296
Title: Emotional Working Memory Training for Veterans With Elevated Trauma-related Symptoms
Brief Title: Emotional Working Memory Training for Veterans With PTSD Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milwaukee VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sadie Larsen, Assistant Professor, Milwaukee VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5134-03
Record Dates: First submitted 2016-05-04; First posted 2016-05-09 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; trauma; working memory; working memory training
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Emotional Working Memory Training (Experimental): Each participant will receive 15 sessions (each lasting 20 minutes) over a 5 week. This will be Internet-based cognitive training based on the adaptive dual n-back paradigm.
  Interventions: Behavioral: Active Emotional Working Memory Training
- Control Working Memory Training (Placebo Comparator): Participants in this condition will receive 15 sessions (each lasting 20 minutes) over a 5-week period. This will also be home-based training over the Internet. This training will be based on a fixed 1-back training program.
  Interventions: Behavioral: Control Working Memory Training

INTERVENTIONS:
Behavioral: Active Emotional Working Memory Training — This training regimen has adapted the existing n-back paradigm, which has been widely used in the field. Training requires participants to shift between visual and auditory information while continually updating their working memory.
  Arms: Active Emotional Working Memory Training
Behavioral: Control Working Memory Training — This training utilized a fixed dual 1-back training paradigm.
  Arms: Control Working Memory Training

SUMMARY:
PTSD is characterized by recurrent intrusion of trauma-related memories and images that cause significant distress and impairment to the affected individuals. The current project aims to examine whether computerized emotional working memory training (eWMT) can help improve working memory capabilities and reduce trauma-related emotional symptoms among individuals with elevated trauma-related symptoms. Participants will be randomly assigned to one of the two computerized training programs. At baseline, post-training, and 1-month follow-up, participants will be assessed with respect to their emotional symptoms and working memory-related cognitive performance. Pending successful outcomes, this study will provide important knowledge that will guide the future efforts to develop an effective, accessible, and cost-efficient intervention program.

DETAILED DESCRIPTION:
PTSD is characterized by recurrent intrusion of trauma-related memories and images that cause significant distress and impairment to the affected individuals. The long-term objective is to develop an effective cognitive treatment program that can reduce such intrusive cognitions observed among individuals who have been exposed to a significant trauma. The specific objective is to examine whether computerized emotional working memory training (eWMT) can help improve working memory capabilities and reduce trauma-related emotional symptoms among individuals with elevated trauma-related symptoms. eWMT is designed to improve the individual's ability to stay focused on the target and filter out irrelevant information from their working memory, which is expected to improve trauma-related emotional symptoms via the improvement of working memory functioning.

Individuals who display elevated trauma symptoms will be randomly assigned to one of two eWMT conditions: (a) adjustable n-back training (i.e., potent working memory training program), and (b) fixed 1-back training (i.e., training that delivers a limited dose). Participants will be blinded to ensure objective assessment of the intervention effects. Before and after the eWMT intervention, all participants will undergo an assessment session that aims to assess each individual's emotional symptoms and working memory-related cognitive performance. Further, following completion of procedure, participants will be invited for a follow-up assessment to assess the long-term effect of training.

The eWMT intervention will be delivered via Internet. Thus, the current intervention is a home-based Internet intervention, which provides an important context for testing and developing a cost-efficient, accessible, and effective intervention program for many individuals suffering from exposure to traumas. Each training session will take about 20 minutes, and all participants in both conditions will receive a total of 15 training sessions. Participants will be guided to complete an average of 3 training sessions every week for a total duration of approximately 5 weeks.

Investigators hypothesize that individuals who undergo the active eWMT will display a greater improvement in overall working memory performance and a greater reduction in trauma-related symptoms, compared to individuals who undergo the less effective control training program. Pending successful outcomes, this study will provide important knowledge that will guide the future efforts to develop an effective, accessible, and cost-efficient intervention program that can reach out to many individuals who suffer from exposure to traumas.

ELIGIBILITY:
Inclusion Criteria:

* Fluently speaks English
* The PTSD Checklist (PCL-5) total score >= 38

Exclusion Criteria:

* No access to a private computer with high-speed Internet that can be used privately.
* Elevated suicidality
* History of psychotic disorders (e.g., schizophrenia)
* Severe substance use disorder (as per DSM-5 criteria)
* History of severe brain injury or organic mental syndrome

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Change in Severity of trauma-related symptoms from baseline to post-training and 1-month follow-up | At baseline, at post-training (after 5 weeks), and at follow-up (1 month from the completion of training)
  PTSD Checklist (PCL-5)

SECONDARY OUTCOMES:
Change in working memory performance from baseline to post-training and 1-month follow-up | At baseline, at post-training (after 5 weeks), and at follow-up (1 month from the completion of training)
  Automated Complex Span Tasks (Oswald et al., 2014). This is a well-validated computerized measure of working memory capacity, including three sub-domains: (1) Operation span, (2) Reading span, and (3) Symmetry span.

OTHER OUTCOMES:
Change in physiological reactivity to the description of one's own traumatic experience from baseline to post-training and 1-month follow-up | At baseline, at post-training (after 5 weeks), and at follow-up (1 month from the completion of training)
  Each participant will be guided to listen to the audiotaped version of his/her own traumatic experience while trying to recollect the event as vividly as possible. Raw ECG signals will be recorded before, during, and after the recollection to measure changes in heart rate variability as an index for emotional regulation and physiological reactivity.

CONTACTS AND LOCATIONS:
Overall Officials: Sadie Larsen, Ph.D., Principal Investigator — Clement J. Zablocki VA Medical Center
Locations (1):
- Clement J. Zablocki VA Medical Center, Milwaukee, Wisconsin, United States